CLINICAL TRIAL: NCT02092571
Title: An Open-Label, Single-Dose, Randomized, 2-Treatment, 2-Period Crossover Pharmacokinetic Study to Evaluate the Bioequivalence of 2 Progesterone Vaginal Rings 20% (w/w) in Postmenopausal Women
Brief Title: A Pharmacokinetic Study to Evaluate the Bioequivalence of 2 Progesterone Vaginal Rings in Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DR201-BE-10021
Record Dates: First submitted 2014-02-28; First posted 2014-03-20 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): 1 ring intravaginal for 7 days, produced from the new process
  Interventions: Drug: Progesterone vaginal ring,
- Treatment B (Experimental): 1 ring intravaginal for 7 days, produced from the legacy process
  Interventions: Drug: Progesterone vaginal ring,

INTERVENTIONS:
Drug: Progesterone vaginal ring, — Participants will be randomized to receive treatments in 1 of 2 treatment sequences (AB or BA)
  Other Names: Treatment A - DR-201, progesterone vaginal ring, 20% (w/w),; 11 mg/day, produced from the NEW process and; Treatment B - DR-201, progesterone vaginal ring, 20% (w/w),; 11 mg/day, produced from the LEGACY process

SUMMARY:
A study to assess the pharmacokinetics of 2 progesterone vaginal rings in postmenopausal women

ELIGIBILITY:
Inclusion:

1. Naturally postmenopausal woman with an intact uterus, 40 to 70 years of age, inclusive.
2. The subject has serum estradiol and FSH levels that are consistent with the subject being postmenopausal.
3. The subject has no clinically significant abnormality findings observed during pelvic, breast, and vaginal examination or based on mammogram and Pap smear evaluations.
4. The subject will agree to be treated with 1 mg/day estradiol oral tablets for at least 28 days before insertion of the first vaginal ring and throughout the study.

Exclusion:

1. The subject has a history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, urologic, gynecologic, immunologic, dermatologic, neurologic, or psychiatric disease.
2. The subject has a history of toxic shock syndrome.
3. The subject has a history of jaundice associated with previous use of oral contraceptives.
4. The subject has contraindications to the use of estrogen or progesterone that include, but are not limited to, the following:

   * known sensitivity to estrogen or progesterone or related drugs
   * known hypersensitivity to study medication ingredients, including FD&C Yellow No. 5 (tartrazine) present in estradiol tablets
   * undiagnosed vaginal bleeding or high risk for endometrial cancer
   * breast mass on examination
   * known, suspected, or family history of estrogen- or progesterone-dependent neoplasia (now or in the past)
5. The subject has low-grade squamous intraepithelial lesion (LSIL) or worse as observed in the Pap smear at screening. Any other abnormal finding on the Pap smear that the investigator considers clinically significant (such as atypical squamous cells cannot exclude high-grade squamous intraepithelial lesion [HSIL; ASC-H], atypical glandular cells [AGC]); or any Pap result that would necessitate further evaluation by biopsy and/or colposcopy.
6. The subject has any abnormal finding or condition deemed clinically significant by the investigator at screening that is a contraindication to the use of progestins, estrogen, or a vaginal ring.
7. The subject has a positive pregnancy test at screening or at any time during the study.
8. Current treatment with progesterone, other progestins, or estrogen (other than estradiol 1-mg tablets, progesterone 200-mg capsules, or medroxyprogesterone acetate 10-mg tablets required for this study purpose).
9. Use of any of the following medications within the time frames noted below before the start of estrogen treatment:

   * vaginal hormonal products (rings, creams, or gels) within 7 days
   * transdermal estrogen alone or estrogen/progestin products within 28 days
   * oral estrogen or progestin therapy within 56 days
   * intrauterine progestin therapy within 56 days
   * progestin implants or estrogen alone injectable drug therapy within 3 months
   * estrogen pellet therapy or progestin injectable therapy within 6 months
10. The subject has a vaginal ultrasonography at screening that confirms an active endometrial lining and/or an endometrial thickness of ≥4 mm.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
baseline-adjusted AUCt | 16 weeks
baseline-adjusted AUC∞ | 16 weeks
baseline-adjusted Cmax | 16 weeks

SECONDARY OUTCOMES:
baseline-adjusted tmax | 16 weeks
baseline-unadjusted AUCt | 16 weeks
baseline-adjusted λz | 16 weeks
baseline-adjusted t½ | 16 weeks
baseline-unadjusted AUC∞ | 16 weeks
baseline-unadjusted Cmax | 16 weeks
baseline-unadjusted tmax | 16 weeks
baseline-unadjusted λz | 16 weeks
baseline-unadjusted t½ | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site 12355, Miami, Florida, United States